CLINICAL TRIAL: NCT00941915
Title: A Phase II Study of Stereotactic Body Radiotherapy (SBRT) for Prostate Cancer Using Continuous Real-time Evaluation of Prostate Motion and IMRT Plan Reoptimization Based on the Anatomy of the Day
Brief Title: Stereotactic Body Radiotherapy (SBRT) for Prostate Cancer
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018266
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer
Keywords: CaP; SBRT; Prostate; ExacTrac; Calypso; IMRT; Radiation; Cancer of Prostate; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Radiotherapy (Experimental): Five fractions of 7.4 Gy each
  Interventions: Radiation: SBRT Prostate

INTERVENTIONS:
Radiation: SBRT Prostate — Five fractions of 7.4 Gy. The total dose will be 37 Gy. A minimum of 36 hours and a maximum of 96 hours should separate each treatment. No more than 3 fractions will be delivered per week. The total duration of treatment will be no shorter than 10 days and no longer than 18 days.
  Other Names: Stereotactic body radiation therapy; External beam radiation therapy

SUMMARY:
The purpose of this study is to evaluate the incidence of urinary and gastrointestinal acute and late side effects in patients treated with stereotactic body radiotherapy (SBRT) to the prostate. Stereotactic radiation therapy is given as five treatments over a 2-3 week period. The prostate is localized and the plan is reoptimized as needed prior to each treatment.

DETAILED DESCRIPTION:
This protocol requires radiation treatments to be performed with a stereotactic technique with the use of a 3-D coordinate system defined by implanted transponders (i.e. Calypso) or use of the ExacTrac system and/or use cone-beam CT (CBCT) with fiducial markers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate within 365 days of study enrollment
* History/physical examination with digital rectal examination of the prostate within 8 weeks prior to study enrollment
* Gleason score less than or equal to 7
* Clinical Stage T1-T2c
* PSA
* less than or = 15 ng/ml prior to start of therapy if Gleason < or = 6 or
* less than or = 10 ng/ml prior to start of therapy if Gleason = 7
* Zubrod Performance Status 0-1
* Age > 40

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years. (Carcinoma in situ of the bladder or oral cavity is permissible)
* Evidence of distant metastases
* Regional lymph node involvement
* Significant urinary obstruction
* Estimated prostate gland > 100 grams
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous hormonal therapy, such as LHRH agonists (e.g. goserelin, leuprolide), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g., DES), or surgical castration (bilateral orchiectomy) or planned concurrent androgen deprivation therapy
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Prosthetic implants in the pelvic region that contain metal or conductive materials (e.g., an artificial hip).
* Severe, active comorbidity

Ages: 40 Years to 82 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R Lee, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Peeters ST, Heemsbergen WD, Koper PC, van Putten WL, Slot A, Dielwart MF, Bonfrer JM, Incrocci L, Lebesque JV. Dose-response in radiotherapy for localized prostate cancer: results of the Dutch multicenter randomized phase III trial comparing 68 Gy of radiotherapy with 78 Gy. J Clin Oncol. 2006 May 1;24(13):1990-6. doi: 10.1200/JCO.2005.05.2530. PMID 16648499
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Madsen BL, Hsi RA, Pham HT, Fowler JF, Esagui L, Corman J. Stereotactic hypofractionated accurate radiotherapy of the prostate (SHARP), 33.5 Gy in five fractions for localized disease: first clinical trial results. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):1099-105. doi: 10.1016/j.ijrobp.2006.10.050. PMID 17336216
- [Result] Boyer MJ, Papagikos MA, Kiteley R, Vujaskovic Z, Wu J, Lee WR. Toxicity and quality of life report of a phase II study of stereotactic body radiotherapy (SBRT) for low and intermediate risk prostate cancer. Radiat Oncol. 2017 Jan 13;12(1):14. doi: 10.1186/s13014-016-0758-8. PMID 28086825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Radiotherapy
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Genitourinary Acute Toxicity
Description: Genitourinary Acute Toxicity is defined as Grade 3 or higher occurring within 90 days from the end of radiation treatment
Time Frame: </= 90 days post radiation treatment, a total of 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 60
Participants
  Grade 1 | 44
  Grade 2 | 15
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

2. Primary Outcome: Number of Participants With Genitourinary Late Toxicity
Description: Genitourinary Late Toxicity is defined as Grade 3 or higher occurring >90 days from the end of radiation treatment
Time Frame: >90 days from the end of treatment, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 60
Participants
  Grade 1 | 22
  Grade 2 | 4
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

3. Primary Outcome: Number of Participants With Gastrointestinal Acute Toxicity
Description: Gastrointestinal Acute Toxicity is defined as Grade 3 or higher occurring within 90 days of the end of radiation treatment
Time Frame: </= 90 days post radiation treatment, a total of 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 60
Participants
  Grade 1 | 19
  Grade 2 | 3
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

4. Primary Outcome: Number of Participants With Gastrointestinal Late Toxicity
Description: Gastrointestinal Late Toxicity is defined as Grade 3 or higher occurring > 90 days from the end of radiation treatment
Time Frame: >90 days from the end of treatment, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 60
Participants
  Grade 1 | 15
  Grade 2 | 5
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

5. Secondary Outcome: Disease Free Survival
Time Frame: 5 yrs
Population: Data not collected.
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life, as Measured by the Expanded Prostate Cancer Index Composite (EPIC-26) Short Form
Description: The EPIC-26 Short Form is a 13-item questionnaire. Scores range from 0-100, with higher scores representing better quality of life.
Time Frame: 3 years post-treatment
Population: Only participants who provided responses for each domain were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiotherapy
Number analyzed (Participants) | 19
score on a scale
  Urinary Domain | 94.1 (14.7)
  Sexual Domain: number analyzed (Participants) | 16
  Sexual Domain | 77.7 (27.6)
  Bowel Domain: number analyzed (Participants) | 17
  Bowel Domain | 90.2 (24.0)
  Hormonal Domain: number analyzed (Participants) | 17
  Hormonal Domain | 94.4 (8.6)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Only Genitourinary and Gastrointestinal adverse events were reported.
Arm/Group | Stereotactic Radiotherapy
All-Cause Mortality (participants affected / at risk) | 4/60
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 51/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiotherapy (N=60)
Proctitis (Gastrointestinal disorders) | 1 (1) — defined as Grade 3 or higher
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiotherapy (N=60)
Diarrhea (Gastrointestinal disorders) | 17 (17)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 4 (4)
Proctitis (Gastrointestinal disorders) | 9 (9)
Rectal hemorrhage (Gastrointestinal disorders) | 14 (14)
Rectal pain (Gastrointestinal disorders) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 51 (51)
Urinary retention (Renal and urinary disorders) | 30 (32)
Urinary tract pain (Renal and urinary disorders) | 22 (22)
Urinary urgency (Renal and urinary disorders) | 28 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT00941915/Prot_SAP_000.pdf